CLINICAL TRIAL: NCT05245747
Title: Vitls Feasibility Physiologic Monitoring
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Vitls Inc. (Industry); American College of Cardiology (Other)
Responsible Party: Principal Investigator, Lori Erickson, Director, Remote Health Solutions, Children's Mercy Hospital Kansas City
Other Study IDs: Study00001853
Record Dates: First submitted 2022-01-19; First posted 2022-02-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Vital Signs; Pediatrics; Remote Monitoring
Keywords: pediatric; physiologic vital signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Vitls Tego Device — The Tégo VSS Sensor is a battery-operated adhesive patch with integrated sensors and wireless transceiver which is worn on the upper body and records heart rate (HR), respiration rate, blood oxygen levels (SpO2), and body temperature. The Tégo VSS Sensor continuously gathers multiparameter physiological data from the person being monitored and then transmits the encrypted data via bi-directional communication to a third-party connectivity relay.
  Other Names: Tego VSS Sensor

SUMMARY:
A single site, cross-sectional, feasibility study will be used to evaluate the feasibility of the collection of physiologic data related to the use of the Vitls Platform in the pediatric (< 2 year of age) congenital heart and general surgery populations in the hospital setting that is using 24 hour a day monitoring for routine care over a 48-hour period. A short questionnaire will be sent electronically for the parent-child dyad feedback after the participating child has worn the device. No data will be available at the time of placement for the Healthcare team and will not replace any routine/standard of care monitoring already in place for this complex population.

DETAILED DESCRIPTION:
After disbursement of information sheet has occurred and verbal parental consent has been obtained, the research staff will determine the initial date of implementation of the Vitls Platform based on need and clinical status. Outcomes will include initiation (first date/time used), persistence (frequency of Tégo and Vitls platform use between first date of use and last date of use and any issues with transfer of data), and feasibility (actual fit with physiologic heart rate, respiratory rate, temperature, and oxygen saturation) compared with standard monitoring data.

After the Tégo sensor has been worn, an electronic REDCap survey for feedback from the parent-child dyad via email or via mobile phone (whichever is the preferred method at enrollment). The researchers will obtain the preferred method of documentation/contact at time of enrollment by the parent entering that into the REDCap. If the child-parent dyad is discharged and a study team member is not available, a link will be sent by the preferred method.

ELIGIBILITY:
Inclusion Criteria:

* • Study participants will be pediatric patients who have undergone cardiac surgery, interventional or diagnostic cardiac catheterizations or former preterm infants undergoing a general surgery procedure at Children's Mercy Kansas City and are currently less than 2 years of age at the time of being approached for participation in this study.

  * Parents of qualifying subjects will also be included in this study.

Exclusion Criteria:

* • Two years of age or older

  * Left sided thoracotomy incision
  * Removal for sternal wound with infection/erythema to site
  * Parents under the age of 18 at the time the study team would approach the family.
  * Infants less than 37 weeks gestation at birth or as determined appropriate by the study team.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Maximum of 50 infants to be enrolled (with the hope to have evaluable data from 20 of these subjects - i.e. this will allow us to account for possible participant attrition, particularly in the beginning of the trial, and the enrollment of up to 25 patients will allow for the learning curve that will have to be overcome by the study team).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Vital sign Heart Rate Feasibility | 90 days
  To evaluate the feasibility of collecting heart rate data with the Vitls Platform
Vital sign Oxygen saturation Feasibility | 90 days
  To evaluate the feasibility of collecting oxygen saturation data with the Vitls Platform
Vital sign Temperature Feasibility | 90 days
  To evaluate the feasibility of collecting temperature data with the Vitls Platform
Vital sign respiratory rate Feasibility | 90 days
  To evaluate the feasibility of collecting respiratory rate data with the Vitls Platform

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erickson, PhD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar N, Akangire G, Sullivan B, Fairchild K, Sampath V. Continuous vital sign analysis for predicting and preventing neonatal diseases in the twenty-first century: big data to the forefront. Pediatr Res. 2020 Jan;87(2):210-220. doi: 10.1038/s41390-019-0527-0. Epub 2019 Aug 4. PMID 31377752
- [Background] Sasangohar F, Davis E, Kash BA, Shah SR. Remote Patient Monitoring and Telemedicine in Neonatal and Pediatric Settings: Scoping Literature Review. J Med Internet Res. 2018 Dec 20;20(12):e295. doi: 10.2196/jmir.9403. PMID 30573451
- See also: Vitls Website — https://www.vitlsinc.com/